CLINICAL TRIAL: NCT00486564
Title: A Phase I Trial of Nifurtimox for Relapsed or Refractory Neuroblastoma
Brief Title: Safety Study of Nifurtimox for Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: St. Louis University (Other)
Responsible Party: Giselle Sholler, MD, University of Vermont
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V0610
Record Dates: First submitted 2007-06-12; First posted 2007-06-14 (Estimated); Last update posted 2009-10-23 (Estimated); Status verified 2009-10

CONDITIONS: Neuroblastoma
Keywords: Treatment; Refractory or Relapsed
MeSH Terms: conditions — Neuroblastoma; Recurrence | interventions — Nifurtimox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nifurtimox — Escalating dose by cohort starting at 20mg/kg/day. PO drug taken TID.

SUMMARY:
There is currently no curative treatment for children with relapsed/refractory neuroblastoma, and for these children the 5 year survival rate is <10%. As such, new therapeutic approaches are needed to treat these children. This Phase 1 clinical trial is specifically designed to test the safety and toxicity of nifurtimox when given in combination with cyclophosphamide and topotecan for the treatment of relapsed and/or refractory neuroblastoma . Prior to study opening, 3 pediatric patients with neuroblastoma have received nifurtimox in combination with this chemotherapy regimen, and all have had significant measurable responses without undue toxicity. These case reports, as well as our in vitro and in vivo investigations into the biologic effect of nifurtimox on neuroblastoma cells has prompted the development of this Phase I study. This Phase I study will involve a dose escalation trial of daily oral nifurtimox alone for one 21 day cycle of therapy, followed by continuation of nifurtimox with the addition of standard doses of cyclophosphamide (5 days) and topotecan (5 days) for 3 additional 21 day cycles. Our primary aim is to evaluate the safety of nifurtimox alone and in combination with these chemotherapy agents in multiply relapsed/refractory patients. Our secondary aim will be to evaluate the pharmacokinetics of nifurtimox as well as treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-21 years at the time of study entry.
2. Diagnosis: Histologic verification of neuroblastoma at original diagnosis or relapse.
3. Disease Status: Refractory or first or multiple relapsed neuroblastoma with measurable disease by radiographic scan (CT or MRI and MIBG), abnormal urinary catecholamine levels, or positive bone marrow biopsy/aspirate. MIBG not required if subject's neuroblastoma is previously determined to not uptake MIBG isotope (not MIBG avid).
4. Current disease state must be one for which there is currently no known curative therapy.
5. A negative urine pregnancy test is required for female participants of child bearing potential (>13 years of age).
6. Patients must have adequate liver function as defined by AST or ALT <10x normal and a bilirubin <1.5mg/dl
7. Informed Consent: All patients and/or legal guardians must sign informed written consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

1. Life expectancy <3 months
2. Investigational Drugs: Patients who are currently receiving another investigational drug.
3. Anti-cancer Agents: Patients who are currently receiving other anticancer agents.
4. Infection: Patients who have an uncontrolled infection.
5. Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study.
6. Patients may not receive bisphosphonates (i.e. Zometa) within 7 days of start of therapy.

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Test the safety of nifurtimox in children with relapsed or refractory neuroblastoma alone and in combination with cyclophosphamide and topotecan. | 3 months

SECONDARY OUTCOMES:
To evaluate the pharmacokinetic profile of nifurtimox alone and in combination with cyclophosphamide and topotecan. | 3 months
To determine the response rate to treatment with nifurtimox combined with cyclophosphamide/topotecan | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Sholler, MD, Study Chair — University of Vermont / Vermont Children's Hospital
Locations (2):
- United States (2):
  - St. Louis University/Cardinal Glennon Childrens Medical Center, St Louis, Missouri
  - University of Vermont/Vermont Children's Hospital, Burlington, Vermont

REFERENCES:
- [Background] Saulnier Sholler GL, Kalkunte S, Greenlaw C, McCarten K, Forman E. Antitumor activity of nifurtimox observed in a patient with neuroblastoma. J Pediatr Hematol Oncol. 2006 Oct;28(10):693-5. doi: 10.1097/01.mph.0000212994.56812.f2. PMID 17023833